CLINICAL TRIAL: NCT06009913
Title: What is More Effective Online Versus Real Time Dental Education
Brief Title: Online Versus Real Time Dental Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Nabil Ahmed Khirat El Hadidi, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 21/8/2023asu
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Educational Problems

STUDY DESIGN:
Intervention Model Description: two group survey 40 students had online teaching 40 students had real time teaching
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: triple blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online teaching (Experimental): Teaching was done completely online
  Interventions: Other: online teaching
- Conventional class room (Active Comparator): Teaching was done completely offline in classroom
  Interventions: Other: In class teaching

INTERVENTIONS:
Other: online teaching — teaching of subject was done using online system only
  Arms: online teaching
Other: In class teaching — subjects were explained in normal class room
  Arms: Conventional class room

SUMMARY:
Through covid period the concept of distant, online and hybrid learning evolved in reaction to lockdown. This hindered the capability of students to receive and practice on patients as they should do. The current study compared data of two classes that had different education systems because of COVID-19. Class 2020 had nearly a complete online teaching of theoretical part, practical and minimal patient interaction. Class 2021 had the opportunity to try both systems because of partial lockdown in 2020 and complete return to work in 2021.

DETAILED DESCRIPTION:
Methodology

Evaluation of the quality of teaching of oral surgery curriculum during the COVID 19 lock down.

The Objective Achieving high quality teaching in similar future situations. The Standards used for evaluation. The course report published by the faculty student's affair section and the students survey.

ETHICS & ENGAGEMENT This data was collected from the course report published by the faculty student's affair section. All students shared in the survey consented that their data can be used and presented for research and audit purposes. All adjunctive research presented in this audit got ethical clearance from the Faculty Ethical Committee.

sample Fourth year students studying oral surgery had online teaching and forty students had real time teaching.

Survey Questions A short five-question survey was used to assess the students overall and was given to 40 students from each class to assess the student's satisfaction with the quality of the education.

The survey questions:

1. Technical skills taught during the academic year were valuable or not.
2. real patients provide higher skills compared to dummies and models
3. Teaching in real classroom is better than teaching through online portal
4. do you prefer introudction of dummies before real time patients
5. Regarding the overall satisfaction by the education system The survey portal had a percentage satisfactory meter. Responses over 50% or equal 50% were considered yes and responses below 50% were considered no.

Statistical assessment:

Chi-square test was used to assess the statistical significance between the results using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* fourth year students attending normally in ain shams university

Exclusion Criteria:

* any student who is repeating or had this course before

Ages: 20 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
effectiveness of online teaching | 3 months
  through a survey 40 students will volunteer for online teaching education survey assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed diaa, Study Chair — Ain shams
Locations (2):
- Egypt (2):
  - Faculty of Dentistry Ain Shams University, Cairo
  - Ain shams University, Cairo

IPD SHARING:
Plan to Share IPD: No
Introduction: Through covid period the concept of distant, online and hybrid learning evolved in reaction to lockdown. This hindered the capability of students to receive and practice on patients as they should do.
  Methodology: The current study compared data of two classes that had different education systems because of COVID-19.

REFERENCES:
- [Result] Haridy R, Abdalla MA, Kaisarly D, Gezawi ME. A cross-sectional multicenter survey on the future of dental education in the era of COVID-19: Alternatives and implications. J Dent Educ. 2021 Apr;85(4):483-493. doi: 10.1002/jdd.12498. Epub 2020 Dec 1. PMID 33263205